CLINICAL TRIAL: NCT06948422
Title: A Master Protocol to Investigate the Efficacy and Safety of Orforglipron Once Daily in Participants With Hypertension and Obesity or Overweight: Randomized, Double-Blind, Placebo-Controlled Trials (ATTAIN-HYPERTENSION)
Brief Title: A Master Protocol for Orforglipron (LY3502970) in Participants With Hypertension and Obesity or Overweight: (ATTAIN-Hypertension Screening)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 27223; J2A-MC-GZPL (Other: Eli Lilly and Company); J2A-MC-GZL1 (Other: Eli Lilly and Company); J2A-MC-GZL2 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orforglipron (GZL1) (Experimental): Participants will receive orforglipron orally or placebo.
  Interventions: Drug: Orforglipron; Drug: Placebo
- Orforglipron (GZL2) (Experimental): Participants will receive orforglipron orally or placebo.
  Interventions: Drug: Orforglipron; Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally.
  Other Names: LY3502970
Drug: Placebo — Administered orally.

SUMMARY:
The GZPL master protocol will support 2 independent studies, J2A-MC-GZL1 (GZL1) and J2A-MC-GZL2 (GZL2). The purpose of this study is to create a framework to evaluate the safety and efficacy of orforglipron for the treatment of hypertension in participants with obesity or overweight.

ELIGIBILITY:
Inclusion Criteria:

* Has systolic blood pressure (SBP) ≥ 140 mmHg and/or diastolic blood pressure (DBP) ≥ 90 mmHg (if DBP criteria alone is met, SBP must be ≥130 mmHg) at screening (Visit 1).
* Has SBP ≥ 140 mmHg and/or DBP ≥ 90 mmHg (if DBP criteria alone is met, SBP must be ≥130 mmHg) at week 0 (Visit 3).
* Untreated for hypertension, or on stable antihypertensive medications ≥ 30 days prior to Visit 1.
* Have a body mass index (BMI) ≥ 25 kg/m².

Exclusion Criteria:

* Has SBP ≥170 mmHg and/or DBP ≥110 mmHg at Visit 1 or at Visit 3.
* Has known secondary causes of hypertension
* Have heart failure with reduced ejection fraction (HFrEF) diagnosis
* Have had any of the following conditions within 90 days prior to screening.

  * hospitalization for hypertension or for congestive heart failure
  * acute coronary syndrome or acute myocardial infarction, or
  * cerebrovascular accident (stroke).
* Have type 1 diabetes (T1D)
* Have acute or chronic hepatitis, including a history of autoimmune hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Allocated to Each ISA | Week -8 to Week 0

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (100):
- United States (30):
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Valley Clinical Trials, Inc., Covina, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Care Access - Brandon, Brandon, Florida
  - Northeast Research Institute - Downtown Office, Jacksonville, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Care Access - St. Petersburg, St. Petersburg, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Rochester Clinical Research, LLC, Rochester, New York
  - Remington-Davis, Inc, Columbus, Ohio
  - PriMED Clinical Research, Dayton, Ohio
  - Advanced Research Institute - Tigard, Tigard, Oregon
  - Care Access - Mauldin, Mauldin, South Carolina
  - Dallas Heart and Vascular Consultants, PA, Duncanville, Texas
  - Texas Institute of Cardiology, PA, McKinney, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
  - Advanced Research Institute, Ogden, Utah
  - Carient Heart & Vascular - Manassas, Manassas, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
  - Eastside Research Associates, Redmond, Washington
- Argentina (8):
  - Instituto Médico Especializado (IME), Buenos Aires
  - CIPREC, Buenos Aires
  - CEMEDIC, Buenos Aires
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - INECO Neurociencias Oroño, Rosario
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario
  - Santa Maria de la Salud Centro Medico, San Isidro
- China (12):
  - Beijing Pinggu District Hospital, Beijing
  - China-Japan Union Hospital, Changchun
  - Changde First People's Hospital, Changde
  - Sichuan Provincial People's Hospital, Chengdu
  - The Second Affiliated Hospital of Chongqing Medical University - Yuzhong Campus, Chongqing
  - Jinan Central Hospital, Jinan
  - Lishui Central Hospital, Lishui
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Siping Central People's Hospital, Siping
  - Wuxi People's Hospital, Wuxi
  - Shaanxi provincial people's hospital, Xi'an
- Czechia (9):
  - Top Moravia Health, Brno
  - Ordinace Rihackovi, s.r.o., Brno
  - CTC Hodonin s.r.o., Hodonín
  - MUDr. Sarka Drinkova, Ledeč nad Sázavou
  - CCR Ostrava s.r.o, Ostrava
  - Diahelp s.r.o, Pardubice V
  - Clinoxus, Prague
  - Angiocentrum Komorany, Prague
  - Praglandia s.r.o, Prague
- Germany (9):
  - Zentrum für klinische Studien Bad Homburg, Bad Homburg
  - FutureMeds GmbH, Berlin
  - Zentrum fur klinische Forschung - Köln, Cologne
  - Hausärztlich-Kardiologisches MVZ am Felsenkeller GmbH/Zentrum für klinische Studien, Dresden
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Medizentrum Essen Borbeck, Essen
  - AmBeNet GmbH, Leipzig
  - Familienmedizinisches Zentrum Radowsky, Leipzig
  - RED-Institut GmbH, Oldenburg
- Greece (6):
  - Athens Medical Center - Psychikon branch, Athens
  - General Hospital of Athens "G. Gennimatas", Athens
  - University Hospital of Ioannina, Ioannina
  - G. Gennimatas General Hospital of Thessaloniki, Thessaloniki
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- India (4):
  - Life Care Hospital and Research Centre, Bangalore
  - All India Institute of Medical Sciences, Bhubaneswar
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
  - Ashirwad Hospital and Research Centre, Ulhasnagar
- Japan (5):
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Fukuwa Clinic, Chūōku
  - Takai Internal Medicine Clinic, Kamakura-shi
  - Mikannohana Clinic, Diabetes, Endocrinology and Metabolism, Matsuyama
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi
- Poland (8):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Centrum Medyczne "Hipokrates" S.C. Elżbieta I Grzegorz Grześk, Bydgoszcz
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - IRMED, Piotrkow Trybunalski
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl
  - Private Practice - Dr. Robert Witek, Tarnów
  - Balsam Medica, Warsaw
  - NZOZ Regionalna Poradnia Diabetologiczna, Wroclaw
- Puerto Rico (2):
  - Dorado Medical Complex, Dorado
  - Puerto Rico Medical Research, Ponce
- Spain (7):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital San Rafael - La Coruña, A Coruña
  - EAP Sardenya, Barcelona
  - EAP Osona Sud - Alt Congost S.L.P, Centelles
  - Complejo Asistencial Universitario de León - Hospital de León, León
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Quiron Infanta Luisa, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/